CLINICAL TRIAL: NCT06881784
Title: RASolve 301: Phase 3 Multicenter, Open Label, Randomized Study of RMC-6236 Versus Docetaxel in Patients With Previously Treated Locally Advanced or Metastatic RAS[MUT] NSCLC
Brief Title: Study of Daraxonrasib (RMC-6236) in Patients With RAS Mutated NSCLC (RASolve 301)
Acronym: RASolve 301
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Revolution Medicines, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMC-6236-301
Record Dates: First submitted 2025-03-10; First posted 2025-03-18 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-11

CONDITIONS: NSCLC (Non-small Cell Lung Cancer); Non-Small Cell Lung Cancer; NSCLC; NSCLC (Non-small Cell Lung Carcinoma); NSCLC (Advanced Non-small Cell Lung Cancer)
Keywords: NSCLC; Non-Small Cell Lung Cancer; Lung Cancer; RAS; KRAS; HRAS; NRAS; RAS Q61 Mutation; RAS G12 Mutation; RAS G13 Mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Masking Description: The central reader of the tumor scans will be masked to the patients' treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- daraxonrasib (Experimental): study drug
  Interventions: Drug: daraxonrasib
- docetaxel (Active Comparator): Patients randomized to the comparator control arm will receive docetaxel as the standard of care therapy.
  Interventions: Drug: docetaxel

INTERVENTIONS:
Drug: daraxonrasib — oral tablets
  Arms: daraxonrasib
Drug: docetaxel — intravenous (IV) infusion
  Arms: docetaxel

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of a novel RAS(ON) inhibitor compared to docetaxel.

DETAILED DESCRIPTION:
This is a global, randomized, open-label, Phase 3 study designed to evaluate whether treatment with daraxonrasib will improve progression free survival (PFS) or overall survival (OS) compared to docetaxel chemotherapy in patients with NSCLC who were previously treated. Patients will be randomized in a 1:1 ratio to receive daraxonrasib or docetaxel chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old and has provided informed consent.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Pathologically confirmed NSCLC, either locally advanced or metastatic, not amenable to curative surgery or radiotherapy.
* Measurable disease per RECIST v1.1.
* Adequate organ function (bone marrow, liver, kidney, coagulation).
* One to two prior lines of therapy including an anti-PD-1/anti-PD(L)-1 agent and platinum-based chemotherapy.
* Documented RAS mutation status, defined as Nonsynonymous mutations in KRAS, NRAS, or HRAS at codons 12, 13, or 61 (G12, G13, or Q61).
* Able to take oral medications.

Exclusion Criteria:

* Prior therapy with direct RAS-targeted therapy or docetaxel.
* Untreated central nervous system (CNS) metastases.
* Medically significant comorbidities (significant cardiovascular disease, lung disease, or impaired GI function).
* Ongoing anticancer therapy.
* Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) per Investigator in the RAS G12X-C population (i.e RAS G12X excluding G12C) | Up to approximately 4 years
  PFS is defined as the time from randomization until disease progression or death from any cause, whichever occurs first. Progression is per response evaluation criteria in solid tumors (RECIST) v1.1 and as assessed by Investigator.
Overall survival (OS) in the RAS G12X-C population | Up to approximately 4 years
  OS is defined as the time from randomization until death from any cause.

SECONDARY OUTCOMES:
PFS in the RAS (MUT) population per Investigator | Up to approximately 4 years
  PFS is defined as time from randomization until disease progression or death from any cause, whichever occurs first. Progression is per RECIST v1.1 as assessed by Investigator.
OS in the RAS (MUT) population | up to approximately 4 years
  OS is defined as time from randomization until death from any cause.
Objective response per Investigator in the RAS (G12X-C) and RAS (MUT) populations | Up to approximately 4 years
  Objective response of partial response (PR) or complete response (CR) per RECIST v1.1 as assessed by Investigator.
PFS per BICR in the RAS (G12X-C) and RAS (MUT) populations | Up to approximately 4 years
  PFS is defined as time from randomization until disease progression or death from any cause, whichever occurs first. Progression is per RECIST v1.1 as assessed by blinded independent central review (BICR).
Objective response per BICR in the RAS (G12X-C) and RAS (MUT) populations | Up to approximately 4 years
  Objective response of PR or CR per RECIST v1.1 as assessed by BICR.
Duration of response (DOR) per Investigator and BICR in the RAS (G12X-C) and RAS (MUT) populations | Up to approximately 4 years
  DOR is defined as time from first evidence of objective response (PR or CR) to disease progression or death due to any cause, whichever occurs first, as assessed by Investigator and by BICR.
Time to response (TTR) per Investigator and per BICR in the RAS (G12X-C) and RAS (MUT) populations | Up to approximately 4 years
  TTR is defined as time from randomization to first evidence of objective response (PR or CR), as assessed by Investigator and by BICR.
Treatment effect on quality of life (QoL) using EORTC QLQ-LC13 In the RAS (G12X-C) and RAS (MUT) populations | Up to approximately 4 years
  Time to deterioration (TTD) in selected symptoms (dyspnea, chest pain, cough) defined as the time from randomization to the first onset of 10 points or more deterioration from baseline in the corresponding symptom scales (dyspnea, chest pain, cough) on European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire LC-13 (EORTC QLQ-LC13).
  Change from baseline on EORTC QLQ-LC13 in symptom scales (dyspnea, cough, chest pain).
Treatment effect on quality of life (QoL) using EORTC QLQ-C30 In the RAS (G12X-C) and RAS (MUT) populations | Up to approximately 4 years
  Change from baseline in global quality of life score from European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTC QLQ-C30) questionnaire.
  Change from baseline on EORTC QLQ-C30 functioning domains (physical role, cognitive, emotional, social).
Safety and tolerability in the RAS (G12X-C) and RAS (MUT) population | Up to approximately 4 years
  Incidence of treatment emergent adverse events (TEAEs), treatment related adverse events (TRAEs), serious adverse events (SAEs), changes in vital signs and clinical laboratory tests.
PK characterization of daraxonrasib In the RAS (MUT) population | Up to approximately 4 years
  Blood concentrations of daraxonrasib over time.

CONTACTS AND LOCATIONS:
Locations (113):
- United States (32):
  - Alabama Oncology, Birmingham, Alabama
  - MemorialCare Long Beach Medical Center, Long Beach, California
  - Yale University, Smillow Cancer Center, New Haven, Connecticut
  - Florida Cancer Specialists & Research Institute - South, Fort Myers, Florida
  - BRCR Global, Plantation, Florida
  - Cancer Care Centers of Breevard, Rockledge, Florida
  - Florida Cancer Specialists & Research Institute - North, St. Petersburg, Florida
  - Cleveland Clinic Martin North, Stuart, Florida
  - Florida Cancer Specialists & Research Institute - East, West Palm Beach, Florida
  - University Cancer and Blood Center, Athens, Georgia
  - Center for Care and Discovery, Chicago, Illinois
  - The University of Kansas Cancer Center, Westwood, Kansas
  - Johns Hopkins University of Medicine, Baltimore, Maryland
  - Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health, Detroit, Michigan
  - Washington University School of Medicine - Siteman Cancer Center, St Louis, Missouri
  - St. Vincent Frontier Cancer Center, Billings, Montana
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center at University of North Carolina, Chapel Hill, North Carolina
  - TriHealth Cancer & Blood Institute Research, Cincinnati, Ohio
  - Taylor Cancer Research Center, Maumee, Ohio
  - Oncology Associates of Oregon PC, Eugene, Oregon
  - SCRI Oncology Partners - Tennessee, Nashville, Tennessee
  - Texas Oncology - South Austin, Austin, Texas
  - Texas Oncology Dallas, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology - Gulf Coast, The Woodlands, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Virginia Cancer Specialists, Fairfax, Virginia
- Australia (4):
  - Blacktown Medical Oncology Research, Blacktown, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Mater Misericordiae Limited, South Brisbane, Queensland
  - Sir Charles Gairdner Hospital, Perth, Western Australia
- Belgium (5):
  - Institut Jules Bordet, Anderlecht, Belgium
  - Grand Hôpital de Charleroi - Les Viviers, Gilly
  - AZ Groeninge, Kortrijk
  - UZ Leuven-Campus Gasthuisberg, Leuven
  - AZ Delta, Roeselare
- France (13):
  - CHU Strasbourg - Nouvel Hôpital Civil, Strasbourg, Bas Rhin
  - Hopital Nord - CHU Marseille, Marseille, Bouches-du-Rhône
  - Institut régional du Cancer de Montpellier, Montpellier, Herault
  - CHU Rennes Hôpital Pontchaillou, Rennes, Ille et Vilaine
  - CHU de Grenoble - Hôpital Albert Michallon, La Tronche, Isere
  - CHU Nantes - Hôpital Guillaume et René Laënnec, Saint-Herblain, Loire Atlantique
  - Institut de Cancerologie de l Ouest, Saint-Herblain, Loire Atlantique
  - Centre Leon Berard, Léon, Lyon
  - Hopital Albert Calmette - CHU Lille, Lille, Nord
  - Hôpital Bichat - Claude Bernard, Paris, Paris
  - Hopital Louis Pradel, Bron, Rhone
  - Centre Hospitalier Intercommunal de Créteil, Créteil, Val de Marne
  - CHU Brest - Hôpital Morvan, Brest
- Germany (2):
  - LKI Lungenfachklinik Immenhausen, Immenhausen, Hesse
  - Universitaetsklinikum Essen, Essen, North Rhine-Westphalia
- Hong Kong United Oncology Centre, Hong Kong, Hong Kong
- Ireland (2):
  - Mater Private Hospital, Dublin, Dublin
  - University Hospital Limerick, Cork, Limerick
- Italy (7):
  - IEO Istituto Europeo di Oncologia, Milan, Milano
  - Azienda Socio Sanitaria Territoriale Niguarda, Milan, Milano
  - Istituto Clinico Humanitas, Rossano, Milano
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli, Napoli
  - Azienda Ospedaliero Universitaria Pisana (Presidio di Cisanello), Pisa, Pisa
  - Istituto Nazionale dei Tumori Regina Elena IRCCS, Roma, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome
- Japan (17):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - Fujita Health University Hospital, Toyoake-shi, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - NHO Shikoku Cancer Center, Matsuyama, Ehime
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Hyogo Cancer Center, Akashi, Hyōgo
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Tohoku University Hospital, Sendai, Miyagi
  - Nara Medical University Hospital, Kashihara-shi, Nara
  - Niigata Cancer Center, Niigata, Niigata
  - Kansai Medical University Hospital, Hirakata-shi, Osaka
  - Kindai University Hospital, Osakasayama-shi, Osaka
  - Shizuoka Cancer Center, Nagaizumi-chō, Shizuoka
  - National Cancer Center Hospital, Chuo Ku, Tokyo
  - Cancer Institute Hospital of JFCR, Koto-Ku, Tokyo
  - Wakayama Medical University Hospital, Wakayama, Wakayama
- Netherlands (5):
  - Amsterdam UMC, Locatie VUMC, Amsterdam, Netherlands
  - Erasmus Medisch Centrum, Rotterdam, Netherlands
  - Antoni van Leeuwenhoek, Amsterdam
  - Maastricht University Medical Center P. Debyelaan 25, Maastricht
  - Radboudumc, Nijmegen
- Poland (3):
  - INSTYTUT GENETYKI I IMMMUNOLOGII GENIM sp. z o.o., Lublin
  - Med-Polonia Sp. z o.o., Poznan
  - Aidport Sp. z o.o., Skorzewo
- Pan American Center for Oncology Trials, San Juan, Puerto Rico, Puerto Rico
- Singapore (2):
  - National University Hospital, Singapore, Singapore
  - National Cancer Centre Singapore, Singapore
- South Korea (6):
  - Ajou University Hospital, Gyeonggi-do, Suwon-si
  - Chungbuk National University Hospital, Cheongju-si
  - Chonnam National University Hwasun Hospital, Hwasun
  - Korea University Anam Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
- Spain (5):
  - Complejo Hospitalario Universitario A Coruña, A Coruña, A Coruña
  - Hospital Universitari Dexeus, Barcelona, Barcelona
  - Hospital Universitario La Paz, Fuencarral-El Pardo, Madrid
  - Hospital Universitario HM Madrid Sanchinarro, Madrid, Madrid
  - Hospital de la Santa Creu i Sant Pau, Barcelona
- Switzerland (3):
  - Universitätsspital Basel, Basel
  - HFR Fribourg/Kantonsspital Fribourg, Fribourg
  - Kantonsspital St. Gallen, Sankt Gallen
- Taiwan (5):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung, Taiwan
  - National Cheng Kung University Hospital, Tainan, Taiwan
  - National Taiwan University Hospital, Taipei, Taiwan
  - Taipei Medical University Hospital, Taipei
  - Chang Gung Medical Foundation Linkou, Taoyuan District